CLINICAL TRIAL: NCT03938896
Title: The Effectiveness of Platelet Rich Plasma in Treatment of Chronic Planter Fasciitis
Brief Title: PRP IN Planter Fascitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: code: MS/15.10.08.
Record Dates: First submitted 2019-05-02; First posted 2019-05-06 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2018-09

CONDITIONS: Chronic Plantar Fasciitis
MeSH Terms: conditions — Fasciitis, Plantar | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- platelet rich plasma (Other): It started with puncture of the vein and taking specific amount of autologous blood from the participantnearly a sample of 20 ml of venous blood (Co AY, 2012).The blood sample was put in a sterile tube containing an anticoagulant as sodium citrate.Then the blood sample wascentrifuged for 15 minutes at 1800 rpmwhich leads to separation of the plasma at the top layer from the packed RBCs at the bottom layer. The RBCs layer is removedthenanother centrifugationwas done at 3500 rpm for 10 minuteswhich leads to formation of a more concentratedplatelet layer after removal of PPP(Anitua et al., 2012).Patients were put in supine position. Betadine was used to disinfect the skin of the heel. 1 ml of local anesthesitic (lidocaine) was injected;then, by the same syringe, 2.5 ml of PRP was injected in the tenderestarea.After extraction of the needle, a bandage was puton the injected area.
  Interventions: Other: platelet rich plasma
- corticosteroid (Other): Patients were put in the supine position. Injection was done usingthe medial technique. Identification of the tenderest point of the heel was done by palpation. Antiseptic solution was used to disinfect the skin overlying theheel. Then1ml of 40 mg methylprednisolone acetate and 1 ml of local anaesthetic as lidocaine 2% were injected into the plantar fascia by a 22gauge needle.
  Interventions: Other: corticosteroid

INTERVENTIONS:
Other: platelet rich plasma — Patients were put in supine position. Betadine was used to disinfect the skin of the heel. 1 ml of local anesthesitic (lidocaine) was injected;then, by the same syringe, 2.5 ml of PRP was injected in the tenderestarea.After extraction of the needle, a bandage was puton the injected area. The patient was kept in the supine position for twentyminutes and then discharged
  Arms: platelet rich plasma
Other: corticosteroid — Patients were put in the supine position. Injection was done usingthe medial technique. Identification of the tenderest point of the heel was done by palpation. Antiseptic solution was used to disinfect the skin overlying theheel. Then1ml of 40 mg methylprednisolone acetate and 1 ml of local anaesthetic as lidocaine 2% were injected into the plantar fascia by a 22gauge needle. After injection, participants were advised to stay sitting without foot movement for 15 minutes
  Arms: corticosteroid

SUMMARY:
The present study was carried out on fifty patients with chronicunilateral PF. Patients were recruited from Outpatient Clinic of Physical medicine, Rheumatology and Rehabilitation at Mansoura University Hospital during the period from January 2016 to September 2016. Patients were classifiedrandomly into two groups:the 1stgroup included 25 patients (20 females and 5 males) treated by local corticosteroid injectionand the 2ndgroup included 25 patients (20 females and 5males) treated by PRP injection.

We obtain an informed written consent from each participant sharing in the study. We take approval on our study by the research board of faculty of medicine, Mansoura University, code: MS/15.10.08.

:

DETAILED DESCRIPTION:
The present study was carried out on fifty patients with chronicunilateral PF. Patients were recruited from Outpatient Clinic of Physical medicine, Rheumatology and Rehabilitation at Mansoura University Hospital during the period from January 2016 to September 2016. Patients were classifiedrandomly into two groups:the 1stgroup included 25 patients (20 females and 5 males) treated by local corticosteroid injectionand the 2ndgroup included 25 patients (20 females and 5males) treated by PRP injection.

We obtain an informed written consent from each participant sharing in the study. We take approval on our study by the research board of faculty of medicine, Mansoura University, code: MS/15.10.08.

All patients were subjected to the following:

1- Complete history taking:

a. Personal history: with special stress on: i. Age and sex. ii. Occupation: occupation which needs prolonged standing is a risk factor for PF.

b. Complaint: Taken in the patient's own words with special stress on disease duration. c. Present history: i. Pain as regard onset, course, duration, provocative factors, relieving factors, limitation of movement and diurnal variation.

ii. History of arthritis and joint affection. iii. History of other systems affections:

* Neurological symptoms: (muscle power and sensation of the lower limbs).
* Eye symptoms: (redness, ulcers and blurred vision).
* Gastrointestinal tract (GIT) symptoms: (diarrhea, heart burn and mucus in the stool).
* Urinary tract (UT) symptoms: (dysuria and frequency).
* Skin affection: (ulcers, erythema, papules and nodules). b. Locomotor system examination:
* Of all joints with special stress on the ankle, subtalar andmidtarsal joint including:

  i. Inspection: swelling, deformity and muscle wasting. ii. Palpation: hotness, tenderness. iii. Range of motion: active and passive.
* Clinical examination of the heel:

  * Inspection of any obvious deformities (pesplanus, pescavus and hallux valgus) and skin changes (redness and swelling).

    1. corticosteroid injection: Patients were put in the supine position. Injection was done usingthe medial technique. Identification of the tenderest point of the heel was done by palpation. Antiseptic solution was used to disinfect the skin overlying theheel. Then1ml of 40 mg methylprednisolone acetate and 1 ml of local anaesthetic as lidocaine 2% were injected into the plantar fascia by a 22gauge needle. After injection, participants were advised to stay sitting without foot movement for 15 minutes (Khan et al., 2014).
    2. PRP injection:

It started with puncture of the vein and taking specific amount of autologous blood from the participantnearly a sample of 20 ml of venous blood (Co AY, 2012).The blood sample was put in a sterile tube containing an anticoagulant as sodium citrate.Then the blood sample wascentrifuged for 15 minutes at 1800 rpmwhich leads to separation of the plasma at the top layer from the packed RBCs at the bottom layer. The RBCs layer is removedthenanother centrifugationwas done at 3500 rpm for 10 minuteswhich leads to formation of a more concentratedplatelet layer after removal of PPP(Anitua et al., 2012).

Patients were put in supine position. Betadine was used to disinfect the skin of the heel. 1 ml of local anesthesitic (lidocaine) was injected;then, by the same syringe, 2.5 ml of PRP was injected in the tenderestarea.After extraction of the needle, a bandage was puton the injected area. The patient was kept in the supine position for twentyminutes and then discharged (Say et al., 2014).

Somepatients may have minimal to moderate discomfort afterinjection that may continue for 7 days because PRP stimulates an inflammatory response. So, to control pain, patients shouldapply ice on the heeland also modify activity as tolerated

ELIGIBILITY:
Inclusion Criteria:

* The study included fifty patients with chronic unilateral PF who were diagnosed by history and physical examination.Patients have heel pain (with VAS more than 50 mm) and tightness after waking upin the morning or after sitting for longperiod. Heel pain will typically improve with movement but maybe increasedatthe end of the day with continuouswalking or standing for a long period.On examining the patients,to avoid placing pressure on the painful heel, patients may walk with their affected foot in an equine position. Palpation of the medial plantar calcaneal region will cause a sharp stabbing pain. Passive ankle/first toe dorsiflexion can cause discomfort in the proxi¬mal plantar fascia(Goff and Crawford, 2011).

Exclusion Criteria:

* Patients with the following conditions were excluded:
* Patients with bilateral heel pain.
* Patients who had received previous local steroid injection.
* Patients who had received NSAIDs within one week.
* Patients having anemia with hemoglobin below 10 gm%, bleeding dyscrasias or thrombocytopenia.
* Patients having earlier injury or surgery to the sole.
* Patients having calcaneal stress fracture, Achilles tendinopathy, tarsal tunnel syndrome or seronegativespondyloarthropathy.
* Patients havingpsychiatric disorders.
* Patients having metabolic or endocrine disease.
* Patients with arthritis of the foot.
* Patients having infections, tumours, vascular abnormalities or neuropathy.
* Patients with hepatic

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
change of pain from base line | immediately before injection,1 month after injection,3 monthes after injection,6 monthes after injection
  VAS is a one-dimensionalmethod used largely in adult patients who also haverheumatic diseases for measuring pain intensity.The VAS score is composed of a continuous linewhich may be a horizontal (HVAS) or vertical (VVAS) line. This line is usually 10 cm (100 mm) in length. To measure the intensity of pain, the score is anchored by "no pain" (0 score) and "pain is as bad as it could be" or "worst imaginable pain"(100 score)on the 100 mm scale. The patient can complete the VAS score by himself. The patientplaces a perpendicular line to the VAS line at the point whichrepresents the intensity of his pain.We can usea ruler to determine the score by measuring the distance (mm) on the 10cm line between the "no pain" anchor and the patient's mark, providing a score range from 0 to 100. According tothe measurement of VAS score in postsurgical

SECONDARY OUTCOMES:
change from base linePlantar fasciitis pain and disability scale (PFPS | immediately before injection,1 month after injection,3 monthes after injection,6 monthes after injection
  The score consists of:
  1. VAS: Rate your pain on a scale of 1 to 100÷ 8.3 = score of _______
  2. How many days a week does pain affect your mobility? (1-7) _____
  3. Is the pain on the surface or deep? ___ Surface = 1, Deep = 3
     Pain description:
  4. Where is your pain located? 0= Toes, 1= Ball of foot, 2= Mid sole, 3= Bottom of Heel
  5. In the past 6 weeks how often have you had pain? 0= Every other week 1= Once a week 2= Once a day 3= Many times a day
  6. How often since the onset of pain, have you been pain free? 0= weeks, 1= days, 2= hours, 3= minutes
  7. How long does the pain last? 0= only when I over exert, 1= pain lasts for less than one hour, 2= pain lasts for one to two hours, 3= pain lasts for more than two hours
  8. In the past 6 weeks what time of day is your pain the worst? (Note this specifically for diagnosis of different problems).
  0= Always the same, 1 = Only in the afternoon, 2 = Both day & night, 3 = Only when you first get up 9-
change from base lineThe modified criteria of the Roles and Maudsley score | immediately before injection,1 month after injection,3 monthes after injection,6 monthes after injection
  Patient satisfaction was assessed using the modified criteria of the Roles and Maudsleyscore. The levels on this scale were as follows:
  * Excellent: no pain, patient satisfied with the treatment outcome and unlimited walking without pain.
  * Good: symptoms substantiallydecreased, patient satisfied with the treatment outcome and ability to walk without pain for >1 hour.
  * Acceptable: symptoms somewhat decreased, pain at a more tolerable level than before treatment and patient slightly satisfied with the treatment outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Reham Magdy Shaat, Al Mansurah, Dakahlia Provence, Egypt